CLINICAL TRIAL: NCT04571918
Title: Arthroscopic Treatment of Massive Rotator Cuff Tears With Debridement and or Biodegradable Spacer: a Prospective Randomized Clinical Trial.
Brief Title: Arthroscopic Treatment of Massive Rotator Cuff Tears With Debridement and Biodegradable Spacer.
Acronym: AMRIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Hannah U. Jahr, Resident in Orthopedic surgery, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/930
Record Dates: First submitted 2020-06-29; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Massive Rotator Cuff Tears
Keywords: Ballon spacer; Biodegradable spacer; Subacromial spacer
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participant and physiotherapist who are responsible for the testing will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Biodegradable spacer (Experimental): Intervention group
  Interventions: Procedure: Biodegradable spacer; Procedure: Debridement and biceps tenotomy
- Group B: control group (Active Comparator): Control group
  Interventions: Procedure: Debridement and biceps tenotomy

INTERVENTIONS:
Procedure: Biodegradable spacer — Implantation of a biodegradable balloon used as a subacromial spacer.
  Arms: Group A: Biodegradable spacer
Procedure: Debridement and biceps tenotomy — Surgery with arthroscopic debridement and biceps tenotomy

SUMMARY:
Massive rotator cuff tears are common in the adult population. It is estimated that about 12 % of adults 60 years of age or older suffer from a rotator cuff injury. About 40 % of these injuries are classified as massive rotator cuff tears (MRCT). MRCT propose a great challenge to the affected patient and its doctor. It is a painful condition with few treatment options.

The study aims to investigate the operative treatment for MRCT with the new treatment option proposed by Senecovic. Insertion of a biodegradable balloon as a subacromial spacer has proven promising results so far. To this date there is only small and non-randomized studies on the subject. AMRIS are planning to do a randomized controlled study where group A is treated with arthroscopic debridement, biceps tenotomy and biodegradable spacer, while group B, the control group are treated with arthroscopic debridement and biceps tenotomy.

DETAILED DESCRIPTION:
The study is designed as a double blinded randomized controlled trial. The physiotherapist responsible for the clinical testing and the patient are both blinded. The surgeon knows which group the patient is in but is not responsible for any of the testing. We will randomize with envelopes perioperatively. The participants are randomized in hence "ballon" or "not ballon". In advance of the randomization the surgeon will evaluate if the patient is candidate for partial suture before randomization. We plan to stratify the patients with partial suture to ensure homogeneity between the groups.

The operation will start with arthroscopic debridement and biceps tenotomy in both groups. The patients are thereby evaluated for partial suture and randomized. The insertion of the subacromial spacer is done at the end of the operation for those patients randomized to the group "balloon". Peroperatively the surgeon will classify the grade of osteoarthritis with Outerbridge classification and the state of the rotator cuff and the long head of the biceps tendon.

Postoperative mobilization will be the following:

* 0-2 weeks: Immobilization in a sling. The participant is advised to do simple exercises for shoulder mobilization. Restriction of movement above shoulder level.
* 2-6 weeks: Free mobilization. Advised to avoid heavy lifting.
* 6-12 weeks: Work on increasing range of motion, gradually introduce weight lifting.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a symptomatic massive rotator cuff tear, with fatty infiltration grade 3 or 4 classified on CT by Goutallier et al, or MRI by Fuchs classification.
* Persistent pain for at least 3 months, with documented failure of conservative treatment
* Age ranging from 60 years of age to 85 years of age

Exclusion Criteria:

* Significant shoulder osteoarthritis in the affected shoulder, Hamada classification >2.
* Total rupture of subscapularis tendon and/or teres minor, classified B and E in the Collins classification.
* Comorbidity to the degree that the patient will not be able to participate in the follow up program.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Constant score | Preop, 6 months, 1 year, 2 years, 5 years, 10 years.
  A well review score that takes several factors in to account: active range of motion, activities of daily living, pain and strength. A person with a normal, healthy shoulder should score 100 points, which is maximum score. Constant score is seen as a relatively objective test, as the testing will be performed by a physiotherapist.

SECONDARY OUTCOMES:
WORC | Preop. Postop: 3 months, 6 months, 1 year, 2 years, 5 years, 10 years
  Western Ontario Rotator Cuff Index is a questionnaire that explores 5 domains: physical symptoms, sports and recreation, work, social function, emotions.
X-ray of the shoulder | Preop. Postop: 1. day, 1 year, 2 years, 5 years, 10 years
  Measure the height from the head of the humerus to the acromion
VAS | Preop. Postop: 3 months, 6 months, 1 year, 2 years, 5 years, 10 years
  Visual analog scale for pain in rest, activity and at night. Scale from 0 til 10.
Eq-5D | Preop. Postop: 3 months, 6 months, 1 year, 2 years, 5 years, 10 years
  Questionaire for daily activity

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Ugletveit Jahr, Cand. med, Study Director — Hospital of southern Norway
Locations (2):
- Norway (2):
  - Hospital of Southern Norway, Arendal, Arendal
  - Oslo university hospital, Oslo

IPD SHARING:
Plan to Share IPD: No
To ensure anonymization of participants, there is no plan to share individual data.